CLINICAL TRIAL: NCT06600529
Title: Evaluation of Combined Photo-Biomodulation At Acupuncture Points, Autologous PRP, and Umbilical Cord-Derived Exosome Therapy in Autism Spectrum Disorder: a Randomized Controlled Trial
Brief Title: Combined Photo-Biomodulation At Acupuncture Points, Autologous PRP, and Umbilical Cord-Derived Exosome Therapy in Autism Spectrum Disorder
Acronym: Biomodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iffat Anwar Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAMC004
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: * Estimated Enrollment: 100 Patients
  * Allocation: Randomized
  * Intervention Model: Parallel Assignment
  * Masking: Single (Participant)
  * Primary Purpose: Treatment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Experimental): Standard Care:
  Procedure: Routine conventional Applied Behavioral Analysis (ABA) management and interventions for ASD, as per current clinical guidelines.
  Interventions: Other: Standard Care (in control arm)
- Experimental Group (Experimental): The Group may be provided with three interventions and then compared with the control group in order to evaluate the effects of the said interventions.
  Interventions: Device: Photo-Biomodulation; Biological: Autologous PRP; Biological: Exosome Therapy

INTERVENTIONS:
Device: Photo-Biomodulation — Application at acupuncture points for 20 seconds each week. using 810nm Laser probe
  Arms: Experimental Group
Biological: Autologous PRP — IV injection of Autologous Plasma Rich Platelets (PRP) on Days 0, 15, 30, and 45.
  Arms: Experimental Group
Biological: Exosome Therapy — IV injection of Umbilical Cord-Derived Exosomes at laser acupuncture points Umbilical Cord-Derived Exosomes
  Arms: Experimental Group
Other: Standard Care (in control arm) — Routine conventional including Applied Behavioral Analysis (ABA) for Autism Spectrum Disorder (ASD)
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of a combination of photo-biomodulation at acupuncture points, autologous platelet-rich plasma (PRP), and umbilical cord-derived exosome therapy in children with Autism Spectrum Disorder (ASD). The study will compare these interventions against standard care to determine their impact on the severity of autism symptoms, as measured by the Childhood Autism Rating Scale (CARS) and other related markers.

DETAILED DESCRIPTION:
The study involves three main interventions:

1. Photo-Biomodulation (PBM): PBM will be performed once a week using an 810nm, 210mW laser probe for 20 seconds at each selected acupuncture point.
2. Autologous Platelet-Rich Plasma (PRP): PRP will be administered at 0 Day, 15 Day, 30 Day, and at 45th Day ADP-derived autologous PRP.
3. Exosome Therapy: Exosomes derived from umbilical cord tissue will be injected intravenously at laser acupuncture points. The PRP-exosome sessions will be repeated at 15 Days, 6 weeks, 12 weeks, and 24 weeks.

The study will run over a period of 6 months, with follow-ups and assessments at each phase. The primary outcome measure will be the change in CARS score, with secondary outcomes including additional ASD markers.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of Autism Spectrum Disorder based on DSM-5 criteria

  * Age 3-12 years
  * Stable on current medications for at least 4 weeks prior to study entry
  * Parents or legal guardians willing to provide informed consent

Exclusion Criteria:

* • Severe comorbid medical conditions

  * Prior stem cell or exosome therapy
  * History of hypersensitivity to any component of the interventions
  * Inability to comply with study procedures

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Change in Childhood Autism Rating Scale (CARS) Score (15-60) | Baseline
  Range of CARS Score 15-29.5: Non-autistic. 30-36.5: Mild to moderate autism. 37-60: Severe autism.
Change in Childhood Autism Rating Scale (CARS) Score (15-60) | 12 Weeks
  Range of CARS Score 15-29.5: Non-autistic. 30-36.5: Mild to moderate autism. 37-60: Severe autism.
Change in Childhood Autism Rating Scale (CARS) Score (15-60) | 6 Months
  Range of CARS Score 15-29.5: Non-autistic. 30-36.5: Mild to moderate autism. 37-60: Severe autism.
Change in Childhood Autism Rating Scale (CARS) Score (15-60) | 1 Year
  Range of CARS Score 15-29.5: Non-autistic. 30-36.5: Mild to moderate autism. 37-60: Severe autism.

SECONDARY OUTCOMES:
Assessment of Social Interaction using Autism Diagnostic Observation Schedule (ADOS) | Baseline
  It have 4 modules each module have 28-30 items each item includes rating 0-3 (0 being normal while 3 specifies severe autism)
Assessment of Social Interaction using Autism Diagnostic Observation Schedule (ADOS) | 12 Weeks
  It have 4 modules each module have 28-30 items each item includes rating 0-3 (0 being normal while 3 specifies severe autism)
Assessment of Social Interaction using Autism Diagnostic Observation Schedule (ADOS) | 6 Months
  It have 4 modules each module have 28-30 items each item includes rating 0-3 (0 being normal while 3 specifies severe autism)
Assessment of Social Interaction using Autism Diagnostic Observation Schedule (ADOS) | 1 Year
  It have 4 modules each module have 28-30 items each item includes rating 0-3 (0 being normal while 3 specifies severe autism)

CONTACTS AND LOCATIONS:
Locations (1):
- Iffat Anwar Medical Complex, Lahore, Punjab Province, Pakistan